CLINICAL TRIAL: NCT06500130
Title: Effects of Liraglutide on Body Surface Gastric Mapping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alimetry (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024 FULL 19945
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Gastroparesis; Functional Dyspepsia; Chronic Nausea and Vomiting Syndrome; Healthy
Keywords: Liraglutide; GLP-1 Receptor Agonist; Gastric Motility; Body Surface Gastric Mapping; Gastric Emptying Breath Test
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Intervention Model Description: This is a Open-label, single site, prospective, proof of concept evaluation of the effect of liraglutide, a NZ-approved daily injectableGLP-1 agonist, on Gastric Alimetry (GA) outputs in up to 20 healthy volunteers. GA will be performed at baseline, after a 12-14 day ascending dose of liraglutide, and after a minimum 5 day washout period.
  This approach directly compares GA within subjects with a gastric-focused pharmacological intervention compared to baseline and after a washout phase. The primary endpoint is a change in GA-RI which isa metric used to define gastric dysrhythmia which is seen in disease states such as neuromuscular disorders and gastroparesis. Since there is no reference standard for GA to compare to, this study will instead allow fulfilment of key plausibility criteria for measuring GA in disease (i.e. inducing symptoms and GA changes in healthy subjects with no previous symptoms.) It will also show that the effects are reversible after stopping the medication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liraglutide Group (Experimental): All study participants will be in this group and will have a total of three body surface gastric mapping tests conducted, pre, during and post liraglutide intervention.
  Interventions: Device: Body Surface Gastric Mapping

INTERVENTIONS:
Device: Body Surface Gastric Mapping — All study participants will be in this group and will have a total of three body surface gastric mapping tests conducted, pre, during and post liraglutide.

SUMMARY:
Aim 1: To investigate, in healthy participants, the effect of liraglutide injection on gastric electrophysiology (as measured by body surface gastric mapping using the Gastric Alimetry device) during an 13-dayramping dose of liraglutide and subsequent washout.

Aim 2: Assessment of effect of liraglutide injection on gastrointestinal symptoms and gut-brain wellbeing (as measured by validated symptom App and Alimetry gut-brain wellness Scale, respectively) during an 13-day ramping dose of liraglutide and subsequent washout.

DETAILED DESCRIPTION:
Globally, more than 40% of persons have a functional gastrointestinal(GI) disorder based on the Rome IV diagnostic questionnaire. These disorders encompass gastroparesis and chronic nausea and vomiting syndromes (CNVS; including chronic unexplained nausea and vomiting(CNV) and cyclic vomiting syndrome (CVS)), functional dyspepsia (FD; chronic indigestion), and post-operative gastric dysfunction. The disorders are linked by the fact that no obvious structural cause for their symptoms can be identified, based on investigations such as endoscopy or imaging. However, there is still a lack of diagnostic biomarkers for these functional disorders. Measuring gastric emptying rate with either scintigraphy or a breath test is the only clinically used test of gastric function; if abnormal the patient is listed as having gastroparesis. However, this test fails to clearly explain the symptom pattern and severity, does not predict response to therapy and changes in the test result do not correlate with evolution of clinical symptoms. There is also substantial crossover in symptoms between functional dyspepsia and gastro-esophageal reflux disease, and differentiating these condition scan be challenging.

GLP-1 analogues cause GI distress and weight loss due to their effect on slowing gastric emptying, inducing satiety or loss of appetite, and thus reducing oral intake. GI symptoms such as nausea, similar to symptoms of gastroparesis, are the most common reason for discontinuation of these drugs. Gastric Alimetry (GA) is a new device which measures gastric electrophysiology. We postulate that GA will show changes in gastric spectral analysis as well as symptoms in healthy volunteers on a once daily injectable GLP-1 analogue, liraglutide.

References:

Sperber AD, Bangdiwala SI, Drossman DA, Ghoshal UC, Simren M, TackJ, Whitehead WE, Dumitrascu DL, Fang X, Fukudo S, Kellow J.Worldwide prevalence and burden of functional gastrointestinaldisorders, results of Rome Foundation Global Study.

Gastroenterology. 2021;160(1):99-114 Pasricha PJ, Grover M, Yates KP,Abell TL, Bernard CE, Koch KL, McCallum RW, Sarosiek I, Kuo B, BulatR, Chen J. Functional dyspepsia and gastroparesis in tertiary care areinterchangeable syndromes with common clinical and pathologicfeatures. Gastroenterology. 2021;160(6):2006-17 Parkman, Henry P.,Daniel S. Rim, Jonathan R. Anolik, Simin Dadparvar, and Alan H. Maurer.2024. "Glucagonlike Peptide-1 Receptor Agonists: The Good, the Bad,and the Ugly-Benefits for Glucose Control and Weight Loss with SideEffects of Delaying Gastric Emptying." Journal of Nuclear MedicineTechnology, January. https://doi.org/10.2967/jnmt.123.266800.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form, AND
* Aged between 18 and 65 years old, AND
* Healthy volunteer with no previous history of gastrointestinal disorders/symptoms
* BMI 22-35

Exclusion Criteria:

1. Confirmed diagnosis of a comorbidity known to affect gastric motility (i.e., Parkinson's Disease, Type 1 or 2 Diabetes).
2. Medications in the last 3 months known to impact gastric motility.
3. Any Gastric Surgery
4. Pregnancy or lactation, determined by pregnancy test at timeof enrolment.
5. Known allergy to adhesives and/or skin sensitivities, or any allergy to liraglutide or any components of the liraglutide/Saxenda formulation, or known hypersensitivity to Spirulina, egg, milk or wheat allergens
6. Use of GLP-1 agonist and/or on regular insulin in the past 3months.
7. History of gastroduodenal dysfunction and/or meets the ROME IV symptom criteria for a gastroduodenal disorder of gut-brain interaction (functional dyspepsia, chronic nausea and vomiting syndrome, cyclic vomiting syndrome, rumination syndrome, cannabinoid hyperemesis syndrome, or a belching disorder).
8. History of peptic ulcer, pancreatitis, cholelithiasis, choledocholithiasis, History of kidney or hepatic dysfunction
9. History of psychiatric disturbance requiring medication in the year before enrolment, any history of suicide attempt or eating disorder
10. History of Type II Diabetes or glucose intolerance (treated or untreated)
11. History of cancer other than basal cell skin cancer, and patients with personal or family history of medullary thyroid carcinoma (MTC) or in patients with multiple endocrine neoplasia syndrome type 2 (MEN 2)
12. History of angioedema or urticaria disorder
13. History of cardiac disorder or arrhythmia
14. Any tobacco, vaping or cannabinoid use in the 30 days prior to study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in overall postprandial BSGM Gastric Alimetry Rhythm Index (GA-RI) on treatment compared to baseline. | 2 weeks
  Change in overall postprandial BSGM Gastric Alimetry Rhythm Index (GA-RI) on treatment compared to baseline.

SECONDARY OUTCOMES:
Change in the following symptoms on treatment compared to baseline | 2 weeks
  GCSI-DD (3 day average, last 3 days on treatment vs 3 days baseline) Alimetry total symptom burden Alimetry individual symptoms
Change in overall postprandial BMI-adjusted amplitude on treatment compared to baseline | 2 weeks
  Change in overall postprandial BMI-adjusted amplitude on treatment compared to baseline
Change in GA-RI on treatment to washout | 1 week
  Change in GA-RI on treatment to washout
Change in BMI-adjusted amplitude on treatment to washout | 1 week
  Change in BMI-adjusted amplitude on treatment to washout
Correlation of total symptom burden with change in GA-RI | 4 weeks
  Correlation of total symptom burden with change in GA-RI
Correlation of total symptom burden with change in BMI-adjusted amplitude | 4 weeks
  Correlation of total symptom burden with change in BMI-adjusted amplitude
Change in gastric emptying half-time on treatment compared to baseline | 2 weeks
  Change in gastric emptying half-time on treatment compared to baseline
Correlation of gastric emptying half-time with GA-RI on treatment | 2 weeks
  Correlation of gastric emptying half-time with GA-RI on treatment
Correlation of gastric emptying half-time with total symptom burden on treatment | 2 weeks
  Correlation of gastric emptying half-time with total symptom burden on treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Alimetry Clinic, Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gastric Alimetry® expands patient phenotyping in gastroduodenal disorders compared to gastric emptying scintigraphy. — http://dx.doi.org/10.14309/ajg.0000000000002528
- See also: Defining and phenotyping gastric abnormalities in long-term type 1 diabetes using a novel body surface gastric mapping device. — http://dx.doi.org/10.1016/j.gastha.2023.08.005